CLINICAL TRIAL: NCT06322628
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of VSA006 Injection in Chinese Adult Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of VSA006 in Chinese NASH Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Visirna Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSA006-2001
Record Dates: First submitted 2023-12-22; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Nash
Keywords: efficacy; safety; HSD17β13
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VSA006 low dose (Experimental)
  Interventions: Drug: VSA006
- VSA006 low dose comparator (Placebo Comparator)
  Interventions: Drug: Placebo
- VSA006 high dose (Experimental)
  Interventions: Drug: VSA006
- VSA006 high dose comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSA006 — every 12 weeks, subcutaneous injections
  Arms: VSA006 high dose; VSA006 low dose
Drug: Placebo — every 12 weeks, subcutaneous injections
  Arms: VSA006 high dose comparator; VSA006 low dose comparator

SUMMARY:
Human genetic studies have shown that loss of function (LOF) mutations in HSD17β13 gene have a protective effect on the progression of alcohol-related and non-alcohol-related liver diseases, such as NASH, without significant adverse phenotypes.

VSA006 is a siRNA drug targeting HSD17β13 mRNA in the liver and reduce the protein level of HSD17β13. Based on phase 1 study results in healthy volunteers and NASH/suspected NASH patients, this phase 2 study is designed to evaluate the efficacy, safety, PK profiles and immunogenicity of VSA006 in Chinese NASH patients.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of 24-35 kg/m2 ;
* NASH patients confirmed by liver histopathology: NAS score is ≥ 4 and CRN fibrosis is F2 or F3 ;
* At screening, ALT is > ULN;
* At screening, the liver fat content measured by MRI-PDFF is ≥ 8%;
* Weight change < 5% at least 3 months prior to screening;
* For patient with T2DM, the hypoglycemic agents and HbA1c is stable

Exclusion Criteria:

* Pregnant or lactating women;
* Previous diagnosis of alcoholic liver disease or hepatitis/liver disease due to other causes;
* Previous or current diagnosis of cirrhosis or decompensated cirrhosis;
* Previous or current diagnosis of hyperthyroidism, hypothyroidism, or other diseases that can lead to fatty degeneration of liver;
* Participants diagnosed with type 1 diabetes, or with unstable type 2 diabetes
* Participants who cannot receive an MRI examination;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving ≥ 1 Stage Improvement in Histological Fibrosis with no Worsening of NASH | At week 52
  No Worsening of NASH is defined as no increase in inflammation, ballooning, or steatosis scores in the NAS score.
Percentage of Participants Achieving NASH Improvement with no Worsening of Fibrosis | At week 52
  NASH Improvement indicates a reduction by at least 2 points in the NAS score, with at least one-point reduction in ballooning without increase in steatosis score.

SECONDARY OUTCOMES:
Compared with placebo, the percentage change in serum alanine aminotransferase (ALT) | At week 24, week 52 and week 82
Compared with placebo, the change in liver fat fraction from baseline and liver fat percentage change from baseline | At week 24 and week 52
  measured by magnetic resonance imaging-proton density fat fraction (MRI-PDFF)
Compared with placebo, the percentage of participants with a > 30% decrease in liver fat fraction from baseline | At week 24 and week 52
  measured by magnetic resonance imaging-proton density fat fraction (MRI-PDFF)
Compared with placebo, the change and percentage change in noninvasive markers of fibrosis from baseline: FIB-4, NAFLD fibrosis score, and AST/PLT ratio index (APRI) | At week 24, week 52 and week 82
Percentage of Participants Achieving NASH Resolution with no Worsening of Fibrosis | At week 52
  NASH resolution was defined as a NAS score of 0-1 for inflammation, 0 for ballooning, and no increase in steatosis score
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and their correlation with VSA006 | Up to week 82
Maximum observed concentration (Cmax) of VSA006 | Pre-dose, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose
Time of maximum concentration of VSA006 (Tmax) | Pre-dose, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose
Area under the concentration-time curve from time zero (pre-dose) to the last quantifiable concentration (AUC0-t) of VSA006 | Pre-dose, 0.5, 1, 2, 4, 8, 12 and 24 hours post dose
anti-drug antibodies (ADAs) of VSA006 | up to week 82

IPD SHARING:
Plan to Share IPD: No